CLINICAL TRIAL: NCT00687531
Title: Open Label, 12-week Clinical Trial to Assess Efficacy, Safety, Treatment Adherence and Quality of Life Impact of Mometasone Furoate Dry Powder 400 mcg Once-daily in Persistent Mild-moderate Asthmatic Patients at Least 12 Years Old
Brief Title: Clinical Trial to Assess Efficacy, Safety, Treatment Adherence and Quality of Life Impact of Mometasone Furoate in Asthmatic Patients (Study P04879)(TERMINATED)
Acronym: APEGO
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P04879
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Results first posted 2011-07-20 (Estimated); Last update posted 2024-05-24 (Actual); Status verified 2022-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Mometasone Furoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mometasone Furoate (Experimental): Mometasone Furoate 400 mcg once daily in the evening through 12 weeks.
  Interventions: Drug: Mometasone Furoate

INTERVENTIONS:
Drug: Mometasone Furoate — Mometasone Furoate 400 mcg once daily, in the evening through 12 weeks.
  Other Names: SCH 32088

SUMMARY:
Open label, 12-week clinical trial to assess efficacy, safety, treatment adherence and Quality of Life impact of Mometasone Furoate dry powder 400 mcg once-daily in persistent mild-moderate asthmatic patients at least 12 years old.

Protocol deviations may have occurred that resulted in quality issues associated with reporting of the data.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate and comply with procedures by signing a written informed consent
* 12 years of age or older of either gender and any race
* Women of childbearing potential (includes women who are less than 1 year postmenopausal and currently are or will become sexually active during the study) must be using or agree to use an acceptable method of birth control unless they are surgically sterilized
* Must understand and be able to adhere to dosing and visit schedules, and agree to record symptom severity scores, PEFR values, medication times, and concomitant medications accurately and consistently in a daily diary.
* Diagnosed history of mild-moderate persistent asthma for at least 12 months.
* FEV1 must be >60% of predicted normal or personal best FEV1 during the last 12 months.
* Using daily inhaled corticosteroids for at least 30 days prior to Screening. In the Screening Visit patients FEV1 should be >= 65% to <= 90% predicted.
* Asthma Symptom Total daily (AM+PM) severity score at Screening Visit should be <= 2.
* For two weeks prior to Screening, subjects must have been on a stable regimen of one of the following twice daily regimen: fluticasone propionate (FP) >= 100 - <= 500 mcg/day; budesonide (BUD) >= 200 - <= 1000mcg/day; beclomethasone dipropionate (BDP) >= 200 - <= 1000 mcg/day; triamcinolone acetonide (TA) >= 400 - <= 2000 mcg/day
* During the inhaled corticosteroid (ICS) Dose Reduction period (max. of 4 weeks; min. of 1 week) of sequential ICS Dose Reduction (approximately 50% reduction in daily dose or discontinue according treatment scheme), subjects must demonstrate a measurable loss of asthma control, with both A) Decreased Lung Function (from the Screening value in absolute FEV1 of >= 10% or >= 220ml OR a decrease in AM PEFR of 25% from the average value for the pre-ICS Dose Reduction period on at least 2 consecutive days out of the last 7 days) AND B) Increased Symptoms (Total AM and PM symptom score of >= 10 out of 24 (using 0-3 scale for each of 4 individual symptoms) on at least 2 days out of the last 7 days OR Increased use of rescue medication from the average value for the pre-ICS Dose Reduction period (one week) of >= 2 puffs on at least 2 days out of the last 7 days)
* Once criterion above have been fulfilled, subjects can be initiated if the FEV1 is 60%-80% predicted
* Subjects must agree to inform their usual treating physicians of their participation in this study

Exclusion Criteria:

* Females who are pregnant or breast-feeding.
* Subjects who have not observed the designated washout periods for any of the prohibited medications
* Subjects who have used any investigational product within 30 days or any antibodies for asthma or allergic rhinitis in the past 90 days prior to enrollment.
* Subjects who have any clinically significant deviation from normal in the physical examination that may interfere with the study evaluations or affect subject safety.
* Subjects who have required systemic steroids within the previous month.
* Subjects who are allergic or have an idiosyncratic reaction to corticosteroids.
* Subjects who have required inpatient hospitalization for asthma control within the previous 3 months, or more than once in the previous 6 months.
* Subjects with clinical evidence of chronic obstructive pulmonary disease or lung diseases other than asthma.
* Subjects who have experienced an upper or lower respiratory tract infection within the previous 2 weeks prior to the Screening Visit.
* Subjects with evidence of clinically significant oropharyngeal candidiasis
* Subjects with any clinically significant immunologic, metabolic, cardiovascular, neurologic, hematologic, gastrointestinal, cerebrovascular, or respiratory disease (other than asthma), or any other disorder which may interfere with the study evaluations or affect subject safety.
* Subjects with a history of drug abuse, antagonistic personality, poor motivation, hypochondriasis, or any other emotional or intellectual problems that are likely to limit the validity of consent to participate in the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2006-11; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mometasone Furoate
Started | 385 (Completed screening procedures)
RECEIVED TREATMENT | 281
Completed | 250
Not Completed | 135
Not completed — Did not meet protocol eligibility | 104
Not completed — Adverse Event | 5
Not completed — Lost to Follow-up | 26

BASELINE CHARACTERISTICS:
Arm/Group | Mometasone Furoate
Number analyzed (Participants) | 281
Age, Customized [Number; unit: participants]
  Between 21 and 30 years | 54
  Between 31 and 40 years | 40
  Between 41 and 50 years | 58
  Between 51 and 60 years | 64
  Between 61 and 70 years | 39
  Between 71 and 80 years | 17
  Between 81 and 90 years | 6
  Not Available to Report | 3
Sex/Gender, Customized [Number; unit: participants]
  Female | 199
  Male | 81
  Not Available to Report | 1

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume in 1 Second (FEV1)
Description: Spirometry was performed to measure FEV1, which is the amount of air the participant is able to exhale in 1 second. Normal values for FEV1 in healthy people depend on age and gender, but values between 80% and 120% of the normal value is considered good. Increased FEV1 indicates improvement in asthma control.
Time Frame: Day 1 and Week 12
Population: study completers (per protocol population)
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Mometasone Furoate
Number analyzed (Participants) | 250
Liters
  Initial (Day 1) | 2.18 (0.75)
  Final (Week 12) | 2.6 (0.83)

2. Secondary Outcome: Morning (AM) and Evening (PM) Peak Expiratory Flow Rate (PEFR)
Description: Participants were to record their daily AM and PM PEFR values in a diary. PEFR can be measured using a peak flow meter that was given to the participant. Normal readings are based on a person's gender, age, and height. A reading of 80 to 100% of the usual or normal peak flow readings indicate that the asthma is under good control. Increased PEFR indicates improvement in asthma control.
Time Frame: Day 1 and Week 12
Population: study completers (per protocol population)
Measure: Mean (Standard Deviation); unit: Liters/minute
Arm/Group | Mometasone Furoate
Number analyzed (Participants) | 250
Liters/minute
  Initial AM (Day 1) | 313.3 (111.2)
  Initial PM (Day 1) | 311.12 (111.2)
  Final AM (Week 12) | 393.3 (144.59)
  Final PM (Week 12) | 395.09 (144.59)

3. Secondary Outcome: Number of Items in the Asthma Quality of Life (QOL) Questionnaire and the General QOL Questionnaire That Had a Significant (Positive) Change From Baseline to Endpoint
Description: Questionnaires consisted of items such as General Health Condition (excellent/very good/good/regular/bad), Difficulty to Breathe (always/almost always/considerable part of time/partially/few amount of time/almost never/never), General Asthma Limitations (completely/a lot/enough to be considered/regular/a few/almost nothing/nothing), etc...
  The questionnaires together consisted of 44 questions, each question with categorical variables as response. A Friedman test was performed to determine the significance of change in samples from baseline to endpoint, for each question.
Time Frame: Day 1 and Week 12
Population: study completers (per protocol population)
Measure: Number; unit: questions
Units Other Than Participants: questions
Arm/Group | Mometasone Furoate
Number analyzed (Participants) | 250
Number analyzed (questions) | 44
questions | 41

4. Secondary Outcome: Morning and Evening Asthma Symptoms Based on a 3 Point Scale (4 Individual Symptoms) and 24 Points (Summed).
Description: The symptoms of cough, chest tightness, wheezing, and shortness of breath were each to be graded on a scale of 0 to 3 with 0 being no symptoms present and 3 being very marked symptoms which was disturbing most of the time. Scores were to have been recorded at 12AM and 12PM for a total of 24 points summed.
Time Frame: Day 1 and Week 12
Population: This analysis was not performed due to missing data at the sites.
Arm/Group | Mometasone Furoate
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Nocturnal Awakenings
Time Frame: Day 1 and Week 12
Population: This analysis was not performed due to missing data at the sites.
Arm/Group | Mometasone Furoate
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Puffs of Salbutamol Used Daily
Time Frame: Day 1 and Week 12
Population: This analysis was not performed due to missing data at the sites.
Arm/Group | Mometasone Furoate
Number analyzed (Participants) | 0

7. Secondary Outcome: Investigator's Assessment of Response to Therapy Based on a 5-point Scale
Description: The investigator will assess the subject's response to therapy by interviewing the subject and comparing the current level of symptoms from baseline. A scale of 1 to 5 will be used with 1 being much improved (AM and PM symptom severety/frequency improve >75% from baseline) and 5 being much worse (AM and PM symptom severity/frequency got more than 75% worse from baseline).
Time Frame: Baseline, Week 12
Population: This analysis was not performed due to missing data at the sites.
Arm/Group | Mometasone Furoate
Number analyzed (Participants) | 0

8. Secondary Outcome: Patient's Assessment of Response to Therapy Based on a 5-point Scale
Description: A scale of 1 to 5 will be used with 1 being much improved (AM and PM symptom severety/frequency improve >75% from baseline) and 5 being much worse (AM and PM symptom severity/frequency got more than 75% worse from baseline).
Time Frame: Baseline, Week 12
Population: This analysis was not performed due to missing data at the sites.
Arm/Group | Mometasone Furoate
Number analyzed (Participants) | 0

9. Secondary Outcome: Number of Participants With One or More Mild, Moderate or Severe Asthma Exacerbations
Description: Exacerbation severity will be characterized based on exacerbation classification from the Global Initiative for Asthma (GINA) workshop 2005 and the National Heart Lung and Blood Institute (NHLBI) asthma guidelines.
Time Frame: Day 1 and Week 12
Population: This analysis was not performed due to missing data at the sites.
Arm/Group | Mometasone Furoate
Number analyzed (Participants) | 0

10. Secondary Outcome: Number of Participants Who Adhered to Treatment
Description: The compliance was measured via medication consumption. In the end of the last week of study (Week 12), a review of the remaining study drug in the initial prescribed Twisthaler device was done. A Twisthaler reading of 0 indicates no study drug left and full compliance.
Time Frame: Day 1 to Week 12
Population: study completers (per protocol population)
Measure: Number; unit: participants
Arm/Group | Mometasone Furoate
Number analyzed (Participants) | 250
participants
  Twisthaler reading 0 (zero) | 196
  Twisthaler reading above zero | 29
  Not specified | 25

11. Secondary Outcome: Number of Participants With Use of Rescue Medication in Each Episode
Time Frame: Day 1 and Week 12
Population: This analysis was not performed due to missing data at the sites.
Units Other Than Participants: episodes
Arm/Group | Mometasone Furoate
Number analyzed (Participants) | 0
Number analyzed (episodes) | 0

ADVERSE EVENTS:
Arm/Group | Mometasone Furoate
Serious Adverse Events (participants affected / at risk) | 0/281
Other Adverse Events (participants affected / at risk) | 0/281

LIMITATIONS AND CAVEATS:
Protocol deviations may have occurred that resulted in quality issues associated with reporting of the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
30 days written notice is required prior to submission of study results for publication/presentation so that Sponsor can review the material to be submitted. Sponsor has the right to review/comment on the material & if the parties have any disagreement concerning the appropriateness of the material, the PI and Sponsor must meet to discuss/resolve any issues/disagreement prior to submission. Interim results of the Study may not be published/presented without prior written consent of Sponsor.